CLINICAL TRIAL: NCT01804101
Title: Liposomal Cytarabine and Daunorubicin (CPX-351) for Adults With Untreated High-Risk MDS and Non-APL AML at High Risk of Treatment-Related Mortality
Brief Title: Liposomal Cytarabine-Daunorubicin CPX-351 in Treating Patients With Untreated Myelodysplastic Syndrome or Acute Myeloid Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Roland Walter, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2642.00; NCI-2013-00481 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2642; 2642.00 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2013-03-01; First posted 2013-03-05 (Estimated); Results first posted 2018-05-25 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-04

CONDITIONS: Acute Biphenotypic Leukemia; Acute Myeloid Leukemia; Myelodysplastic Syndrome; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — CPX-351; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (lower-dose liposomal cytarabine-daunorubicin CPX-351) (Experimental): INDUCTION/RE-INDUCTION: Patients receive lower-dose liposomal cytarabine-daunorubicin CPX-351 IV over 90 minutes on days 1, 3, and 5. Treatment repeats every 40 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients achieving CR or CRp continue on to consolidation.
  CONSOLIDATION: Patients receive lower-dose liposomal cytarabine-daunorubicin CPX-351 IV over 90 minutes on days 1 and 3. Treatment repeats every 40 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Liposomal Cytarabine-Daunorubicin CPX-351
- Arm II (closed to accrual effective 4/21/14) (Experimental): INDUCTION/RE-INDUCTION: Patients receive higher-dose liposomal cytarabine-daunorubicin CPX-351 IV over 90 minutes on days 1, 3, and 5. Treatment repeats every 40 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients achieving CR or CRp continue on to consolidation.
  CONSOLIDATION: Patients receive higher-dose liposomal cytarabine-daunorubicin CPX-351 IV over 90 minutes on days 1 and 3. Treatment repeats every 40 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Liposomal Cytarabine-Daunorubicin CPX-351

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Liposomal Cytarabine-Daunorubicin CPX-351 — Given IV
  Other Names: CPX-351; Cytarabine-Daunorubicin Liposome for Injection; Liposomal AraC-Daunorubicin CPX-351

SUMMARY:
This randomized clinical trial studies liposomal cytarabine-daunorubicin CPX-351 in treating patients with untreated myelodysplastic syndrome or acute myeloid leukemia. Drugs used in chemotherapy, such as liposomal cytarabine-daunorubicin CPX-351, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Estimate whether the 32 units/m^2 or the 64 units/m^2 or both dose levels of CPX-351 (liposomal cytarabine-daunorubicin CPX-351) are likely to improve treatment-related mortality (TRM) rate while keeping the complete remission (CR) rate constant in patients with untreated high-risk myelodysplastic syndrome (MDS) or non-acute promyelocytic leukemia (APL) acute myeloid leukemia (AML) at high risk of TRM.

SECONDARY OBJECTIVES:

I. Describe the CR/CR with incomplete platelet count recovery (CRp) rate after up to 4 cycles of induction/re-induction therapy.

II. Describe the event-free survival, disease-free survival, and overall survival of patients who achieve CR/CRp.

III. Estimate the frequency and severity of regimen-associated toxicities.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I:

INDUCTION/RE-INDUCTION: Patients receive lower-dose liposomal cytarabine-daunorubicin CPX-351 intravenously (IV) over 90 minutes on days 1, 3, and 5. Treatment repeats every 40 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients achieving CR or CRp continue on to consolidation.

CONSOLIDATION: Patients receive lower-dose liposomal cytarabine-daunorubicin CPX-351 IV over 90 minutes on days 1 and 3. Treatment repeats every 40 days for 4 courses in the absence of disease progression or unacceptable toxicity.

ARM II: (closed to accrual effective 4/21/14) INDUCTION/RE-INDUCTION: Patients receive higher-dose liposomal cytarabine-daunorubicin CPX-351 IV over 90 minutes on days 1, 3, and 5. Treatment repeats every 40 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients achieving CR or CRp continue on to consolidation.

CONSOLIDATION: Patients receive higher-dose liposomal cytarabine-daunorubicin CPX-351 IV over 90 minutes on days 1 and 3. Treatment repeats every 40 days for 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of untreated "high-risk" MDS (>= 10% blasts) or AML other than acute promyelocytic leukemia (APL) with t(15;17)(q22;q12) or variants according to the 2008 World Health Organization (WHO) classification; patients with biphenotypic AML are eligible; outside diagnostic material is acceptable as long as peripheral blood and/or bone marrow slides are reviewed at the study institution and cytogenetic/molecular information is available

  * Prior hydroxyurea for AML is permitted but should be discontinued prior to start of CPX-351 treatment
  * Azacitidine, decitabine, lenalidomide, and growth factors are permitted for low-risk MDS (< 10% blasts); all treatments for MDS should be discontinued prior to start of CPX-351 treatment
* Treatment-related mortality (TRM) score >= 13.1 as calculated with simplified model
* Bilirubin < 2.0 mg/mL x upper limit of normal; this requirement reflects the excretion of CPX-351 by the liver
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) < 4.0 x upper limit of normal; this requirement reflects the excretion of CPX-351 by the liver
* Left ventricular ejection fraction (LVEF) >= 40%, assessed within 28 days prior to registration, e.g. by multi gated acquisition (MUGA) scan or echocardiography, or other appropriate diagnostic modality
* Patients with symptoms/signs of hyperleukocytosis or white blood cell (WBC) > 100,000/uL can be treated with leukapheresis prior to enrollment
* Provide signed written informed consent

Exclusion Criteria:

* Refractory/relapsing blast crisis of chronic myelogenous leukemia (CML)
* Concomitant illness associated with a likely survival of < 1 year
* Active systemic fungal, bacterial, viral, or other infection, unless under treatment with anti-microbials and controlled/stable, as defined as being afebrile and hemodynamically stable for 24-48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-05-07 (Actual); Primary Completion 2017-01-10 (Actual); Study Completion 2017-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roland Walter, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (2):
- United States (2):
  - Stanford Cancer Institute, Palo Alto, California
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Lower-dose CPX-351): INDUCTION/RE-INDUCTION: Patients receive lower-dose liposomal cytarabine-daunorubicin CPX-351 IV over 90 minutes on days 1, 3, and 5. Treatment repeats every 40 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients achieving CR or CRp continue on to consolidation.
  CONSOLIDATION: Patients receive lower-dose liposomal cytarabine-daunorubicin CPX-351 IV over 90 minutes on days 1 and 3. Treatment repeats every 40 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Correlative studies
  Liposomal Cytarabine-Daunorubicin CPX-351: Given IV
- Arm II (Higher Dose COX-351): INDUCTION/RE-INDUCTION: Patients receive higher-dose liposomal cytarabine-daunorubicin CPX-351 IV over 90 minutes on days 1, 3, and 5. Treatment repeats every 40 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients achieving CR or CRp continue on to consolidation.
  CONSOLIDATION: Patients receive higher-dose liposomal cytarabine-daunorubicin CPX-351 IV over 90 minutes on days 1 and 3. Treatment repeats every 40 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Correlative studies
  Liposomal Cytarabine-Daunorubicin CPX-351: Given IV
Period: Overall Study
Arm/Group | Arm I (Lower-dose CPX-351) | Arm II (Higher Dose COX-351)
Started | 38 | 10
Completed | 38 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm I (Lower-dose Liposomal Cytarabine-daunorubicin CPX-351): INDUCTION/RE-INDUCTION: Patients receive lower-dose liposomal cytarabine-daunorubicin CPX-351 IV over 90 minutes on days 1, 3, and 5. Treatment repeats every 40 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients achieving CR or CRp continue on to consolidation.
  CONSOLIDATION: Patients receive lower-dose liposomal cytarabine-daunorubicin CPX-351 IV over 90 minutes on days 1 and 3. Treatment repeats every 40 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Correlative studies
  Liposomal Cytarabine-Daunorubicin CPX-351: Given IV
- Arm II (Closed to Accrual Effective 4/21/14): INDUCTION/RE-INDUCTION: Patients receive higher-dose liposomal cytarabine-daunorubicin CPX-351 IV over 90 minutes on days 1, 3, and 5. Treatment repeats every 40 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients achieving CR or CRp continue on to consolidation.
  CONSOLIDATION: Patients receive higher-dose liposomal cytarabine-daunorubicin CPX-351 IV over 90 minutes on days 1 and 3. Treatment repeats every 40 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Correlative studies
  Liposomal Cytarabine-Daunorubicin CPX-351: Given IV
- Total: Total of all reporting groups
Arm/Group | Arm I (Lower-dose Liposomal Cytarabine-daunorubicin CPX-351) | Arm II (Closed to Accrual Effective 4/21/14) | Total
Number analyzed (Participants) | 38 | 10 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 2 | 12
  >=65 years | 28 | 8 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 3 | 16
  Male | 25 | 7 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 38 | 10 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 3 | 0 | 3
  Black or African American | 0 | 0 | 0
  White | 35 | 10 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38 | 10 | 48

OUTCOME MEASURES:

1. Primary Outcome: Treatment-related Mortality Rate. (TRM)
Description: Estimate whether the 32 units/m2 or the 64 units/m2 or both dose levels of CPX-351 are likely to improve treatment-related mortality (TRM) rate while keeping the CR rate constant in patients with untreated high-risk MDS or non-APL AML at high risk of TRM.
Time Frame: Up to 1 month after completion of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Lower-dose Liposomal Cytarabine-daunorubicin CPX-351) | Arm II (Closed to Accrual Effective 4/21/14)
Number analyzed (Participants) | 38 | 10
Participants | 6 | 2

2. Secondary Outcome: Overall Remission Rate (CR+CRp)
Description: Overall Remission Rate for the CR/CR with incomplete platelet count recovery (CRp) rate after up to 4 cycles of induction/re-induction therapy.
Time Frame: Up to day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Lower-dose CPX-351) | Arm II (Higher Dose COX-351)
Number analyzed (Participants) | 38 | 10
Participants | 10 | 1

ADVERSE EVENTS:
Time Frame: 3 years
Description: SAE reporting per our institution, is if it's related and unexpected. None of our AE's met this criteria per protocol. AE's are were review by study coordinator and PI threw medical records and outside records from patients other physicians.
Arm/Group | Arm I (Lower-dose Liposomal Cytarabine-daunorubicin CPX-351) | Arm II (Closed to Accrual Effective 4/21/14)
All-Cause Mortality (participants affected / at risk) | 10/38 | 5/10
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/10
Other Adverse Events (participants affected / at risk) | 38/38 | 10/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Lower-dose Liposomal Cytarabine-daunorubicin CPX-351) (N=38) | Arm II (Closed to Accrual Effective 4/21/14) (N=10)
Neutroprenic Fever (Infections and infestations) | 5 (5) | 2 (2)
Increased Creatinine (Endocrine disorders) | 3 (3) | 0 (0)
epistaxis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
PICC Line infection (Infections and infestations) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (5) | 0 (0)
Fatigue (General disorders) | 8 (8) | 2 (2)
Neutropenia (Infections and infestations) | 9 (9) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (7) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Nausea (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
hypoxemia (Infections and infestations) | 2 (2) | 1 (1)
Edema (General disorders) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No